CLINICAL TRIAL: NCT02972398
Title: N-Acetyl Cysteine add-on to Antidepressant Medication in Therapy Refractory Major Depressive Disorder Patients With Increased Inflammatory Activity
Brief Title: N-Acetyl Cysteine Supplementation in Therapy Refractory Major Depressive Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAC-2015-TJAH
Record Dates: First submitted 2016-11-12; First posted 2016-11-23 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2021-10

CONDITIONS: Major Depressive Disorders
Keywords: treatment resistant depression; N-Acetyl Cysteine; inflammation mediators; oxidative stress; brain imaging
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC group (Experimental): Participants of "NAC group" receive 1000 mg NAC twice daily for 12 weeks as add-on to either a selective serotonin reuptake inhibitor (SSRI) or a serotonin and noradrenalin reuptake inhibitor (SNRI)
  Interventions: Drug: N-acetylcysteine
- Placebo group (Placebo Comparator): Participants of "Placebo group" receive placebo matched with NAC twice daily for 12 weeks as add-on to either a selective serotonin reuptake inhibitor (SSRI) or a serotonin and noradrenalin reuptake inhibitor (SNRI)
  Interventions: Drug: placebo comparator of N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Participants of interventional group receive 1000mg N-acetylcysteine twice daily for 12 weeks.
  Other Names: YiWeiShi
  Arms: NAC group
Drug: placebo comparator of N-acetylcysteine — Participants of placebo group receive placebo comparator matching with N-acetylcysteine twice daily for 12 weeks.
  Arms: Placebo group

SUMMARY:
The aim of this study is to evaluate the efficacy of N-acetylcysteine (NAC) add-on to antidepressant medication in treating patients who do not relieve during standard antidepressant treatment for 6 weeks at least. Meanwhile, secondary outcomes will include changes in some biomarkers and on specifically local brain activity (functional Magnetic Resonance Imaging, fMRI) and white matter integrity (Diffusion Tensor Imaging, DTI). The hypothesis of this study is that NAC has positive effects on refractory major depressive disorder patients with increased inflammatory activity.

DETAILED DESCRIPTION:
It's a double-blind randomised placebo controlled antidepressant augmentation study with 12-week treatment and 8-week follow up. Its purpose is to investigate antidepressant efficacy and safety of NAC in patients with treatment resistant depression (TRD) defined as insufficient response to 1 or more antidepressants given for at least 6 weeks and in an adequate dose, displaying increased peripheral inflammatory activity and moderate to severe depression. Apart from studying the effects of NAC on depression severity, the secondary outcomes are to examine a range of biomarkers related to potentially important underlying mechanisms such as oxidative stress and inflammatory activity and to evaluate the effects on brain functioning (fMRI) and on white matter integrity (DTI). Scale assessments are performed in the week preceding initiation of treatment, during the treatment period, at the end of the treatment period and at 8-week follow up. Neuro-imaging is performed before the treatment starts and in week 12, before the study medication is terminated. Collection of blood and morning urine only takes place at three time points, in the week preceding initiation of treatment, closely before tapering off the study medication and at the end of 8-week follow up. This study is hoped to show that NAC perform positive effects on those aspects mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* a current episode of MDD diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR) diagnosed with SCID
* an age between 18 and 65 years
* a total score of HAMD-17 ≥ 17
* a CRP level between 0.85 and 10 mg/L (The CRP range is based on literature values for mild to moderate chronic inflammation, while values > 10 mg/L point at acute inflammation. A pilot study at the Tianjin Hospital (n=62) indicated that approximately one third of all patients with MDD will have CRP values within this range). insufficient response to 1 or more antidepressants given for at least 6 weeks and in an adequate dose during the current episode
* stable dose of the current antidepressant drug for at least 2 weeks prior to initiation of the study
* Patients are allowed to use benzodiazepines (BZD) to relieve anxiety during the first phase of antidepressant treatment (Anding Hospital protocol). Benzodiazepines may also be prescribed because of sleeping problems during the trial. BZD use will be recorded at all assessments during the trial and after follow-up.
* Patients are compliant with treatment according to the judgement of the treating clinician.
* Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods during the study. Clinical patients always get a pregnancy test before start of treatment.
* Participant or guardian has to sign informed consent. The patients' guardians will sign the informed consent on behalf of the participants when the capacity of participants to consent is compromised.

Exclusion Criteria:

* A history of manic episode
* Use of mood stabilizer
* Use of antipsychotic medication with more than half of the maximum dosage suggested in the instruction
* History of substance abuse or dependence
* An allergic reaction to NAC or any component of the preparation
* Severe somatic diseases that might interfere with regular antidepressant treatment including conditions such as kidney and liver failure, uncontrolled hypertension, cardiovascular, cerebrovascular and pulmonary disease, thyroid disease, diabetes, epilepsy and asthma.
* Use of anti-inflammatory medication for longer than 7 days in the last two months preceding the trial
* Use of immunosuppressive medication such as oral steroid hormones
* History of chronic infection, such as Tuberculosis, AIDS, hepatitis
* CRP value > 10 mg/L
* Women in pregnancy or lactation period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The change from baseline Hamilton Depression Rating Scale (HAMD)-17 items at week2,4,6,8,10,and 12. | baseline, Week 2,4,6,8,10, and 12
  The main objective is to investigate whether daily oral NAC administration in addition to regular treatment with an antidepressant will alleviate the severity of MDD symptoms as measured with the HAMD-17 after 12 weeks of treatment compared to placebo addition, and we also look at other time points, such as week 2,4,6,8,and 10.

SECONDARY OUTCOMES:
The change from baseline HAMD-17 items at week14,16,18,and 20. | baseline, Week 14,16,18,and 20.
  We also look at whether daily oral NAC treatment will still have measurable effects on HAMD-17 score at 8 weeks follow-up after discontinuation of NAC treatment.
The effects of augmentation treatment with NAC on scores in Beck Anxiety Inventory (BAI) | baseline, Week 4,8,12,16,and 20.
The effects of augmentation treatment with NAC on scores in Inventory of Depressive Symptoms-Self-Rated (IDS-SR) | baseline, Week 4,8,12,16,and 20.
The effects of augmentation treatment with NAC on scores in WHO Disability Assessment Schedule Ⅱ (WHODAS-Ⅱ) | baseline, Week 4,8,12,16,and 20.
The effects of augmentation treatment with NAC on scores in Montreal Cognitive Assessment (MoCA) | baseline, Week 4,8,12,16,and 20.
The effects of augmentation treatment with NAC on local brain activity (fMRI and DTI) | baseline, the end of week 12.
The effects of augmentation treatment with NAC on a range of biomarkers representing the alleged underlying pathophysiological mechanisms | baseline, the end of the week 12 and 20
  biomarkers associated with inflammation, oxidative stress, and neurogenesis in sample of serum and urine.
Assessments the side effects measured with Checklist of 52 Somatic Items (CSI) | baseline, Week 4,8,12,16,and 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang C, Bosker FJ, Li J, Schoevers RA. N-acetylcysteine as add-on to antidepressant medication in therapy refractory major depressive disorder patients with increased inflammatory activity: study protocol of a double-blind randomized placebo-controlled trial. BMC Psychiatry. 2018 Sep 4;18(1):279. doi: 10.1186/s12888-018-1845-1. PMID 30176835